CLINICAL TRIAL: NCT05681442
Title: Beta-lactam Intermittent Versus Continuous Infusion and Combination Antibiotic Therapy in Sepsis
Acronym: BICCS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180596
Record Dates: First submitted 2022-11-21; First posted 2023-01-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: The study will be a prospective multicentre, randomized, open-label comparative continuous vs. intermittent pivotal βL antibiotic infusion strategies and combination vs. monotherapy trial conducted with a 2X2 factorial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- continuous infusion dosing of a pivotal AND AG infusion for 5 days (Experimental): continuous infusion dosing of a pivotal βL-AB (CID group) AND AG infusion for 5 days (long duration) as appropriate combination therapy (ACT group)
  Interventions: Drug: continuous pivotal βL-AB; Drug: AG infusion for 5 days
- intermittent infusion dosing of a pivotal βL-AB ND AG infusion for 5 days (Experimental): intermittent infusion dosing of a pivotal βL-AB (IID = control group) AND AG infusion for 5 days (long duration) as appropriate combination therapy (ACT = group)
  Interventions: Drug: intermittent pivotal βL-AB; Drug: AG infusion for 5 days
- continuous infusion dosing of a pivotal βL-AB AND AG infusion at most 1 dose (Experimental): continuous infusion dosing of a pivotal βL-AB (CID group) AND AG infusion at most 1 dose (AMT group )
  Interventions: Drug: continuous pivotal βL-AB; Drug: AG infusion most 1 dose
- intermittent infusion dosing of a pivotal βL-AB AND AG infusion at most 1 dose (Experimental): intermittent infusion dosing of a pivotal βL-AB (IID = group) AND AG infusion at most 1 dose (AMT group)
  Interventions: Drug: intermittent pivotal βL-AB; Drug: AG infusion most 1 dose

INTERVENTIONS:
Drug: continuous pivotal βL-AB — continuous pivotal βL-AB
  Other Names: CID group
  Arms: continuous infusion dosing of a pivotal AND AG infusion for 5 days; continuous infusion dosing of a pivotal βL-AB AND AG infusion at most 1 dose
Drug: intermittent pivotal βL-AB — intermittent pivotal βL-AB (IID = control group)
  Other Names: IID control group
  Arms: intermittent infusion dosing of a pivotal βL-AB AND AG infusion at most 1 dose; intermittent infusion dosing of a pivotal βL-AB ND AG infusion for 5 days
Drug: AG infusion most 1 dose — AG infusion most 1 dose (AMT group )
  Other Names: AMT group
  Arms: continuous infusion dosing of a pivotal βL-AB AND AG infusion at most 1 dose; intermittent infusion dosing of a pivotal βL-AB AND AG infusion at most 1 dose
Drug: AG infusion for 5 days — AG infusion for 5 days (ACT Group)
  Other Names: ACT Group
  Arms: continuous infusion dosing of a pivotal AND AG infusion for 5 days; intermittent infusion dosing of a pivotal βL-AB ND AG infusion for 5 days

SUMMARY:
Patients hospitalized in ICU with sepsis (infection with life-threatening organ dysfunction according to sepsis 3.0 definitions) or septic shock presumably due to MDR-GNB (multidrug resistant Gram-negative bacteria). The study will be a prospective multicentre, randomized, open-label comparative continuous vs. intermittent pivotal βL (Beta Lactamine) antibiotic infusion strategies and combination vs. monotherapy trial conducted with a 2X2 factorial design.

DETAILED DESCRIPTION:
The study will be a prospective multicentre, randomized, open-label comparative continuous vs. intermittent pivotal βL antibiotic infusion strategies and combination vs. monotherapy trial conducted with a 2X2 factorial design.

Patients will be randomized to one of four of the following treatment groups in a 1:1:1:1 ratio. Randomization will be stratified on the centre and the initial βL administered (meropenem versus other) to receive (i) βL antibiotic either as a continuous infusion: CID group or as intermittent infusion: IID group, and (ii) either at most 1 dose (short duration) : AMT group or 5 days (long duration) : ACT group of aminoglycoside

* Arm A: continuous infusion dosing of a pivotal βL-AB (Antibiotics) (CID group) AND AG (Aminoglycoside) infusion for 5 days (long duration) as appropriate combination therapy (ACT group)
* Arm B: intermittent infusion dosing of a pivotal βL-AB (IID = control group) AND AG infusion for 5 days (long duration) as appropriate combination therapy (ACT = group)
* Arm C: continuous infusion dosing of a pivotal βL-AB (CID group) AND AG infusion at most 1 dose (AMT group)
* Arm D: intermittent infusion dosing of a pivotal βL-AB (IID = group) AND AG infusion at most 1 dose (AMT group)

The primary objective of the study is to compare the 30-day mortality of patients with hospital-acquired sepsis in the ICU according to the mode of administration of the pivotal βL antibiotic (CID group vs. IID group).

The primary endpoint is the mortality rate at day 30 between CID and IID groups while the Co-primary objective is to compare the MAKE 30 (Major Adverse Kidney Events within 30 days) between patients that will receive an appropriate monotherapy with βL (AMT group) or an appropriate combination therapy with βL and 5 days of AG (ACT group).

moreover, The co-primary criterion is the percentage of patients with a MAKE 30, i.e. when patients met one of the following criteria within day 30: in-hospital mortality, receipt of renal replacement therapy (RRT) or persistent renal dysfunction (discharge serum creatinine/baseline serum creatinine ≥200%) between AMT and ACT groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* Hospital-acquired sepsis (according to sepsis 3.0 definitions) :

  * Patient hospitalized for more than 48 hours OR Patient discharged less than 48 hours ago
  * AND sepsis diagnosed within the last 24 hours
* One of the following risk factors for gram negative multidrug resistant pathogens:

  * Prior intravenous antibiotic use within 7 days prior to sepsis onset with the exception of antibiotic effective only against Gram-positive bacteria, penicillin A and macrolides
  * Prolonged hospital stay (≥ 15 days of hospitalization) within 3 months prior to sepsis onset Prolonged mechanical ventilation (≥ 5 days on mechanical ventilation) within 3 months prior to sepsis onset
  * Patients with indwelling devices (dialysis access lines, intravascular lines, urinary catheter, endotracheal or tracheostomy tube, gastrostomy or jejunostomy feeding tube)
  * Patients known to be infected, colonized or carriers of MDR gram negative bacteria within 3 months prior to sepsis onset
  * Exposure to an antibiotic (amoxicillin-clavulanic acid, C2G, C3G, fluoroquinolones) within 3 months prior to sepsis onset
  * A trip abroad to known geographical areas at risk (in particular the Indian subcontinent, South-East Asia, the Middle East and North Africa, the Mediterranean Basin) within 3 months prior to sepsis onset
  * A functional or organic abnormality of the urinary tract in case of urinary tract infection.
* Appropriate bacteriological sampling performed before starting antimicrobial therapy
* Expected stay in ICU of more than 3 days

Exclusion Criteria:

* A priori known resistance to all the proposed beta-lactams or to amikacin
* Need for extrarenal treatment at inclusion according to the criteria of Gaudry et al.
* Known hypersensitivity to ceftazidime, piperacillin-tazobactam, cefepime, meropenem, ceftazidime-avibactam, ceftazolane-avibactam or to any of the excipients included in the corresponding pharmaceutical drugs,
* Known hypersensitivity to any cephalosporin antibacterial agent,
* Know hypersentitivity to any penem antibacterial agent,
* Severe known hypersensitivity (eg, anaphylactic reaction, severe skin reaction) to any other beta-lactam antibiotic (eg, penicillins or monobactam ) or to any of its excipients.
* Known contraindication to the aminoglycoside family including

  * Hypersensitivity to the active substance, to any aminoglycoside antibacterial agent or to any of the excipients included in the corresponding pharmaceutical drugs,
  * Cirrhosis of grades B and C according to the Child-Pugh classification.
  * Myasthenia gravis.
  * Simultaneous administration of another aminoglycoside
  * Association with ataluren
* Non-complicated urinary tract infection (corresponding to a positive ECBU not responsible for sepsis)
* Bone marrow transplant or chemotherapy-induced neutropenia
* Infections for which long-term antibiotic treatment > 8 days is strongly recommended (i.e., infective endocarditis, osteoarticular infections, anterior mediastinitis after cardiac surgery, hepatic or cerebral abscesses, chronic prostatitis for instance
* Presence of antibiotic therapyfor the new sepsis before randomisation: (> 2 doses of antibiotics or > 16h for continuous infusion
* Limitation of life support (comfort care applied only) at the time of screening
* Enrolment to another interventional drug study
* Pregnancy or breastfeeding
* Subject deprived of freedom, subject under a legal protective measure
* Non affiliation to any health insurance system
* Refusal to participate to the study (patient or legal representative or family member or close relative if present)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare the 30-day mortality of patients with hospital-acquired sepsis in the ICU | 30 days after acquiring sepsis
  the primary objective is to compare the 30-day mortality of patients with hospital-acquired sepsis in the ICU according to the mode of administration of the pivotal βL antibiotic (CID group vs. IID group).

SECONDARY OUTCOMES:
New carriage, colonization or infection with one of the following BMR-GNB: at days 3, 7 and 30: | days 3,7and 30
  Percentage of patients with new carriage of MDR-GNB(taking into account all clinical samples and rectal surveillance swabs performed routinely each week),i.e one of the following ticarcillin-resistant Pseudomonas aeruginosa,Acinetobacter baumannii,or Stenotrophomonas maltophilia; extended-spectrum β-lactam-producing Entero bacteriaceae;high-concentration cephalosporinase producing AmpC Enterobacteriaceae;
30 day mortality in patient with proven Gram-negative infection | 30 days after inclusion
  Mortality rate at day 30 in patients with proven GNI
30 day mortality in patient with proven non-fermentative GNI | 30 days after inclusion
  Mortality rate at day 30 in patients with proven non-fermentative GNI,
30 day mortality in patient with proven GNI for which the minimum inhibitory concentration (MIC) of the βL used were higher to the breakpoints according to the European committee on Antimicrobial Susceptibility Testing (EUCAST). | 30 days after inclusion
  Mortality rate at day 30 in patients with proven GNI for which the MIC of the βL used were higher to the accepted break-points
30-day mortality in patients that received non-carbapenem-βL | 30 days after inclusion
  Mortality rate at day 30 in patients that received non-carbapenem-βL
30-day clinical recovery | 30 days after inclusion
  Clinical recovery at day 30 defined as admission clinical symptom resolved
30-day clinical recovery | 30 days after inclusion
  Clinical recovery at day 30 defined as admission organ failures resolved with persistence of admission clinical symptoms and time to clinical recovery
PK-PD (pharmacokinetic-pharmacodynamic) target attainment | at day 1, i.e. 24 hours after the loading dose and at day 3, i.e. 72 hours after the loading dose
  PK-PD target attainment rate evaluated as a dichotomous variable
  o For βL (trough or plateau concentration according to randomization group), at day 1, i.e. 24 hours after the loading dose and at day 3, i.e. 72 hours after the loading dose
  § Target attainment scored "Yes" if measured drug concentration exceeded greater than four times to the causative pathogen MIC as 100% fT > 4*MIC
PK-PD (pharmacokinetic-pharmacodynamic) target attainment | 30 min after the end of the first infusion dose (CMAX)
  For AG, 30 min after the end of the first infusion dose (CMAX)
  § Target attainment scored "Yes" if measured drug concentration to causative pathogen MIC ratio is greater than 12 as CMAX/MIC > 12
Superinfection (primary infection site) or new infection (different infection site) at day 30 due to a GNB resistant to the βL administered at inclusion | 30 days after inclusion
  Percentage of patients with superinfection or new nosocomial infection with GNB resistant to the βL administered at inclusion until day 30
Microbiological failure persistence of the same microorganism at the same site at end-of-therapy (EOT) or within 7 days after EOT. | 7 days after inclusion
  Percentage of patients for whom the microorganism is still recovered in bacterial culture from the initial infected site at EOT or within 7 days after EOT
New carriage, colonization or infection with Pseudomonas aeruginosa not susceptible to the βL administered at days 3, 7 and 30 | 30 days after inclusion
  Percentage of patients with new carriage colonization or infection with Pseudomonas aeruginosa not susceptible to the βL administered until day 30
Duration of organ failure between day 1 and day 30 | day 1 and day 30
  Organ failures assessed by AUCSOFA and its organ components measured between day 1 and day 30
Length of ICU and hospital stays | 30 days after inclusion
  Length of ICU and hospital stays until day 30
Occurrence of adverse events at day 30 | 30 days after inclusion
  Percentage of patients with encephalopathy (delay between inclusion and 2 RASS scores = -1 in a row) or renal failure at discharge (RRT or persistent renal dysfunction) until day 30
180-day mortality | 180 days after inclusion
  Mortality rate at day 180

CONTACTS AND LOCATIONS:
Overall Officials: Aline DECHANET, Study Chair — Assistance Publique - Hôpitaux de Paris (AP-HP)
Locations (28):
- France (28):
  - Médecine intensive - réanimation - CHU Amiens-Picardie, Amiens
  - Réanimation polyvalente - CH d'Argenteuil - Hôpital Victor Dupuy, Argenteuil
  - Réanimation polyvalente - CH Avignon, Avignon
  - Médecine intensive - réanimation - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - Médecine intensive - réanimation - Ambroise Paré, Boulogne-Billancourt
  - Médecine intensive - réanimation - CHU Gabriel Montpied, Clermont-Ferrand
  - Anesthésie - Réanimation - Beaujon, Clichy
  - Réanimation polyvalente/Surveillance continue - CH Sud Essonne-Etampes, Étampes
  - Médecine intensive - réanimation-Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Médecine intensive - réanimation - CHU Grenoble-Alpes Hôpital Michallon, La Tronche
  - Réanimation polyvalente - CH de Versailles - Hôpital André Mignot, Le Chesnay
  - Réanimation Médico Chirurgicale & USC - CH Le Mans, Le Mans
  - Médecine Intensive Réanimation - Hôpital Croix Rousse, Lyon
  - Médecine intensive - réanimation - HCL - Edouard Herriot, Lyon
  - Réanimation polyvalente - CHR Metz-Thionville - Hôpital de Mercy, Metz
  - Médecine intensive - réanimation - CHU Montpellier - Hôpital Lapeyronie, Montpellier
  - Réanimation Chirurgicale - Saint Eloi, Montpellier
  - Médecine Intensive Réanimation - Pasteur 2, Nice
  - Médecine intensive - réanimation - CHU Nice - Hôpital Archet, Nice
  - Médecine intensive - réanimation, Orléans
  - Anesthésie - Réanimation - CHU Orléans, Orléans
  - Médecine intensive et réanimation infectieuse - Bichat, Paris
  - Réanimation chirurgicale - Bichat, Paris
  - Institut Mutualiste du Montsouris, Paris
  - Médecine intensive - réanimation - CHU Poitiers - Site de la Milétrie, Poitiers
  - Médecine intensive et réanimation polyvalente 6 CHU de Reims - Hôpital Robert Debré, Reims
  - Médecine intensive - réanimation-CH St Denis - Hôpital Delafontaine, Saint-Denis
  - Médecine intensive - réanimation - CHU de Strasbourg - Nouvel Hôpital Civil, Strasbourg

IPD SHARING:
Plan to Share IPD: No